CLINICAL TRIAL: NCT06110520
Title: Violet Light for Treatment of Myopia
Brief Title: Violet Light for the Suppression of Myopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0289
Record Dates: First submitted 2023-06-13; First posted 2023-10-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Phototherapy
Keywords: Myopia; Violet Light
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Three single groups:
  1. Violet + / Lens + Lamp emits violet light and subjects are either wearing no refractive correction or wearing CR-39 lenses that completely transmit violet light.
  2. Violet + / Lens - Lamp emits violet light and subjects are wearing violet-filtering glasses that block out violet light from reaching their eyes.
  3. Violet - / Lens - Lamp does not violet light and subjects are wearing CR-39 lenses that completely transmit violet light.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized into one of three study groups. The patient, their caregiver, and the investigator will be masked to their treatment group. The study coordinator will organize the patients study treatment and assist in any issues that arise to keep both the patient and investigator masked at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Violet + / Lens + (Experimental): Subjects use a violet light emitting lamp (device intervention - minimally invasive as it's simply a source of light) with CR-39 lenses for their refractive correction. The lamp introduces violet light (Violet +) and the CR-39 lenses allow for the transmission of violet light through the lenses (Lens +).
  Interventions: Device: Violet Light Lamp
- Violet + / Lens - (Experimental): Subjects use a violet light emitting lamp (device intervention - minimally invasive as it's simply a source of light) with polycarbonate lenses for their refractive correction. The lamp introduces violet light (Violet +) while the polycarbonate lenses block the transmission of violet light through the lenses (Lens -).
  Interventions: Device: Violet Light Lamp
- Violet - / Lens + (Placebo Comparator): Subjects use a lamp with NO violet light (Violet -) with CR-39 lenses for their refractive correction. CR-39 lenses allow for the transmission of violet light through the lenses (Lens +).
  Interventions: Device: White Light Lamp

INTERVENTIONS:
Device: Violet Light Lamp — Medical grade lamps with Violet LEDs enabled
  Arms: Violet + / Lens +; Violet + / Lens -
Device: White Light Lamp — Standard bedside lamp with standard 4000K LED light bulb.
  Arms: Violet - / Lens +

SUMMARY:
The study explores the suppression of myopia via violet light.

DETAILED DESCRIPTION:
The study uses violet light-emitting lamps as the variable and regular, white light lamps as the control in assessing whether violet light, especially during over periods of dawn and dusk could help suppress the progression of myopia in developing children.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between 5 to <13 years old.
* Diagnosis of Myopia (ICD-10-CM Diagnosis

Code H52.13) with refractive error:

1. Myopia -1.00D to -6.00D spherical equivalent (SE) in both eyes
2. Astigmatism <=1.50D in both eyes
3. Anisometropia <=1.00D SE • Relocation outside of the CCHMC area within the next 12 months is not anticipated.

Exclusion Criteria:

Current or previous myopia treatment with atropine, pirenzepine, or other antimuscarinic agents

* Current or previous use of bifocals, progressive addition lenses, or multi-focal contact lenses
* Current or previous use of orthoK, rigid gas permeable, or other contact lenses being used to reduce myopia progression
* Current or prior history of manifest strabismus, amblyopia, or nystagmus
* Abnormality of cornea, lens, central retina, iris, or ciliary body
* Prior eyelid, strabismus, intraocular, or refractive surgery
* Down syndrome or cerebral palsy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Axial Length | Measured at baseline, and 12 months.
  Measurement of the distance between anterior cornea and retina via IOL Master in millimeters.
Refractive Error | Measured at baseline, and 12 months.
  The measurement of power eye measured in diopters.
Visual Acuity | Measured at baseline, and 12 months.
  The measurement of how well a person can see letters at a specific distance, measured in logMAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT06110520/Prot_000.pdf